CLINICAL TRIAL: NCT00002974
Title: A Phase II Study of Whole Blood Hyperthermia and Ice Chemotherapy in Sarcoma Patients
Brief Title: Whole-Body Hyperthermia Plus Chemotherapy in Treating Patients With Advanced Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065489; WCCC-CO-9672; NCI-G97-1217
Record Dates: First submitted 1999-11-01; First posted 2004-03-30 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2011-05

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Carboplatin; Etoposide; Ifosfamide; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carboplatin
Drug: etoposide
Drug: ifosfamide
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Hyperthermia therapy kills tumor cells by heating them to several degrees above body temperature. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with whole-body hyperthermia may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of whole-body hyperthermia plus combination chemotherapy in treating patients who have advanced sarcoma that is metastatic or that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the combination of 41.8 degrees Celsius whole body hyperthermia (WBH) and ifosfamide/carboplatin/etoposide (ICE) chemotherapy in patients with advanced sarcoma. II. Assess the efficacy of this combination of therapy. III. Assess the clinical toxicity of WBH and ICE in these patients. IV. Obtain pilot data on the effect of WBH and ICE on cytokine induction in these patients.

OUTLINE: Treatment of whole body hyperthermia (WBH) and ifosfamide/carboplatin/etoposide (ICE) is given every 3-4 weeks. On day 1 of the treatment, ifosfamide is administered intravenously over 60 minutes at the beginning of hyperthermia. Carboplatin is administered intravenously over 20 minutes while at the maximum temperature. Etoposide is administered intravenously over 60 minutes while receiving hyperthermia and on day 2 and 3 after hyperthermia. Patient disease status is reevaluated after 2 courses. If there is no disease progression, treatment continues for a maximum of 4 courses.

PROJECTED ACCRUAL: Approximately 17-34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced sarcoma that is metastatic or incurable surgically Evaluable or measurable disease Must be refractory to all known forms of effective therapy No CNS tumor involvement No major liver involvement (more than 33% replacement of liver by tumor)

PATIENT CHARACTERISTICS: Age: 18-65 Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC greater than 3,000/mm3 Absolute granulocyte count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Alkaline phosphatase no greater than 3 times normal SGOT no greater than 3 times normal Protein no less than 15% below lower limit of normal Renal: BUN less than 30 mg/dL Creatinine less than 1.5 mg/dL OR Creatinine clearance no less than 60 mL/min Calcium no greater than 11.0 mg/dL Sodium 130-150 mmol/L Potassium 3.0-5.0 mmol/L Cardiovascular: No organic heart disease - coronary artery disease - history of angina - history of dysrhythmia requiring ongoing medical intervention - uncontrolled hypertension - patients that require beta blockers - congestive heart failure Neurologic: No tumor involvement of CNS No moderate or severe peripheral neuropathy No history of severe emotional instability by psychiatric history Pulmonary: FEV1 at least 60% of predicted Maximum voluntary volume at least 60% of predicted Partial pressure of oxygen at least 60 OR Oxygen saturation at least 90% Other: No history of secondary primary cancer which conceivably could be active No active nonmalignant gastric and/or duodenal ulcer No serious infection requiring hospitalization within the previous 14 days No history of hepatitis related to general anesthesia No history of allergy to lidocaine or related compound No development of malignant hyperthermia after general anesthesia No unexplained persistent fever Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 8 weeks since nitrosoureas (e.g., CCNU, BCNU, mitomycin) At least 4 weeks since any other chemotherapy Recovered from all toxic effects Endocrine therapy: Not specified Radiotherapy: No prior irradiation of more than 25% of the marrow Surgery: Not specified Other: No concurrent nonsteroidal anti-inflammatory agents or aspirin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 1996-07; Primary Completion 2001-07 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. I. Robins, MD, PhD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States